CLINICAL TRIAL: NCT05003466
Title: A Randomized, Double-blind, Placebo-controlled Phase Ⅱ Clinical Study to Evaluate the Safety and Immunogenicity of Inactivated SARS-CoV-2 Vaccine (Vero Cells) in Healthy Population Aged 3 to 17 Years
Brief Title: Study of Inactivated SARS-CoV-2 Vaccine (Vero Cells) in Healthy Population Aged 3 to 17 Years(COVID-19)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen Kangtai Biological Products Co., LTD (Industry)
Collaborators: Beijing Minhai Biotechnology Co., Ltd (Industry); Hunan Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020L001-2B
Record Dates: First submitted 2021-08-10; First posted 2021-08-12 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- candidate vaccine (Experimental)
  Interventions: Biological: SARS-CoV-2 Vaccine (Vero Cells), Inactivated
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 Vaccine (Vero Cells), Inactivated — 2 doses of SARS-CoV-2 Vaccine (Vero Cells), Inactivated with a 28-day interval constitute a primary immunization course. The third dose on 6 months after primary course is the booster dose.
  Administer as an intramuscular injection into the lateral deltoid of the upper arm.
  Arms: candidate vaccine
Biological: Placebo — 2 doses of Placebo should be administered as an intramuscular injection into the lateral deltoid of the upper arm with a 28-day interval.
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blinded, and placebo controlled phase Ⅱ clinical trial of the SARS-CoV-2 inactivated vaccine to evaluate the safety and immunogenicity of the experimental vaccine in healthy population aged 3 to 17 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy residents aged 3 to 17 years at the time of consent
* Subjects and/or their guardian agree to sign the informed consent forms voluntarily.
* Be able to comply with study requirements/procedures.
* Axillary temperature ≤ 37.0℃

Exclusion Criteria:

* Within 14 days before vaccination, subjects have been abroad and to villages/communities experienced COVID-19 epidemics, and in contact with COVID-19 cases or suspected cases. Subjects are under isolation observation, or living in the villages/communities with COVID-19 cases or suspected cases;
* Confirmed cases, suspected cases or asymptomatic cases with COVID-19 (refer to Information System of China Disease Prevention and Control);
* Subjects with history of SARS virus infection by self-reported;
* Positive in throat swab through RT-PCR;
* History of vaccination of various COVID-19 vaccines or positive in SARS-CoV-2 antibody test;
* Positive urine pregnancy test for females with menarche
* History of severe allergic reactions (such as acute anaphylaxis, urticaria, skin eczema, dyspnea, angioneurotic edema or abdominal pain) or allergy to known composition of inactivated SARS-CoV-2 vaccine;
* History or family history of convulsion, epilepsy, encephalopathy or mental illness;
* Subjects with congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.;
* Subjects with known or suspected diseases include: severe respiratory diseases, severe cardiovascular diseases, severe liver and kidney diseases, drug-uncontrollable hypertension, diabetic complications, malignant tumors, various acute diseases or acute onset of chronic diseases;
* Diagnosed with congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases;
* History of coagulation dysfunction (e.g. Coagulation factor deficiency, coagulation disease);
* Subjects receiving anti-TB treatment;
* Subjects receiving other research drugs within 6 months before vaccination;
* Subjects receiving immunotherapy or inhibitor therapy within 3 months (consistently oral or infusion for more than 14 days);
* Subjects receiving blood products within 3 months before administration;
* Subjects vaccinated with live attenuated vaccine within 14 days before vaccination;
* Subjects vaccinated with other vaccine within 7 days before vaccination;
* The researchers shall judge the other conditions which might be not in compliance with the requirements of this clinical trial.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate of SARS-CoV-2 neutralizing antibody | 28 days post full primary immunization course
Geometric mean titer of SARS-CoV-2 neutralizing antibody | 28 days post full primary immunization course

SECONDARY OUTCOMES:
Incidence of adverse reactions/events | 0-28 days after each vaccination
Serious Adverse Events (SAE) | within 12 months post full primary immunization course and the booster dose respectively
Seroconversion rate of SARS-CoV-2 IgG binding antibody | 28 days post full primary immunization course
Geometric mean titer of SARS-CoV-2 IgG binding antibody | 28 days, 3 months, 6 months and 12 months post full primary immunization course
Geometric mean titer of SARS-CoV-2 IgG binding antibody | 28 days, 3 months, 6 months and 12 months after the booster dose
Geometric mean titer of SARS-CoV-2 neutralizing antibody | 3 months, 6 months and 12 months post full primary immunization course
Geometric mean titer of SARS-CoV-2 neutralizing antibody | 28 days, 3 months, 6 months and 12 months after the booster dose
Seropositive rate of SARS-CoV-2 neutralizing antibody | 3 months, 6 months and 12 months post full primary immunization course
Seropositive rate of SARS-CoV-2 neutralizing antibody | 28 days, 3 months, 6 months and 12 months after the booster dose
Seropositive rate of SARS-CoV-2 IgG binding antibody | 3 months, 6 months and 12 months post full primary immunization course
Seropositive rate of SARS-CoV-2 IgG binding antibody | 28 days, 3 months, 6 months and 12 months after the booster dose

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Provincial Center for Diseases Control and Prevention, Changsha, Hunan, China

REFERENCES:
- [Derived] Liu J, Huang B, Li G, Huang T, Wang D, Zhang L, Deng Y, Chang X, Liu Y, Li W, Zhang S, Huang W, Tan W, Gao L. Immunogenicity and Safety of a SARS-CoV-2 Inactivated Vaccine KCONVAC in Chinese Children: Randomized, Double-blind, Placebo-controlled Phase 1 and 2 Trials. Pediatr Infect Dis J. 2023 Dec 1;42(12):1136-1142. doi: 10.1097/INF.0000000000004085. Epub 2023 Sep 4. PMID 37967148